CLINICAL TRIAL: NCT02038530
Title: D-dimer Testing, Tailored to Clinical Pretest Probability, to Minimize Initial and Follow-up Ultrasound Imaging in Suspected Deep Vein Thrombosis: A Management Study
Brief Title: The Designer D-dimer Deep Vein Thrombosis Diagnosis (4D) Study
Acronym: 4D
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: OCOG-2013-4D
Record Dates: First submitted 2014-01-13; First posted 2014-01-16 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Suspected Deep Vein Thrombosis
Keywords: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- No Ultrasound: Low Clinical Pretest Probability and D-dimer < 1000 ug/L; Moderate Clinical Pretest Probability and D-dimer < 500 ug/L
- Ultrasound Required: Low Clinical Pretest Probability and D-dimer 1000 - 3000 ug/L; Moderate Clinical Pretest Probability and D-dimer 500 - 3000 ug/L; High Clinical Pretest Probability

SUMMARY:
This is a cohort study that will assess a new diagnostic management strategy for suspected Deep Vein Thrombosis in outpatients.The new diagnostic strategy is designed to reduce the use of ultrasound testing on the day of presentation, and reduce repeat ultrasound testing a week after an initial normal test.

DETAILED DESCRIPTION:
This is a prospective, multicentre, cohort study that will assess a new diagnostic management strategy for suspected Deep Vein Thrombosis in outpatients. The new diagnostic strategy is designed to reduce the use of ultrasound testing on the day of presentation, and reduce repeat ultrasound testing a week after an initial normal test. Less ultrasound testing will be performed because: i) more patients will have deep vein thrombosis excluded by combinations of Clinical Pretest Probability and D-dimer results on the day of presentation; and, ii) in those who still need an ultrasound, a repeat ultrasound a week after a normal result will only be performed if the D-dimer result is markedly abnormal at initial presentation. The safety of this management strategy will be established by demonstrating a very low rate of proximal Deep Vein Thrombosis or Pulmonary Embolism during 90 days follow-up in patients who had anticoagulant therapy withheld in response to negative diagnostic testing. Diagnostic test utilization will be assessed. All clinical outcomes will be adjudicated by a central independent adjudication committee that will be blind to initial D-dimer measurements and patient management.

ELIGIBILITY:
Inclusion Criteria:

1) Consecutive outpatients (i.e. non-hospitalized patients) with clinically suspected Deep Vein Thrombosis.

Exclusion Criteria:

1. Age less than 18 years.
2. Treated with full-dose anticoagulation for ≥ 24 hours before D-dimer was measured.
3. D-dimer level known before Clinical Pretest Probability documented.
4. Ultrasound of the leg performed before Clinical Pretest Probability was documented
5. Ultrasound was or will be performed in a patient with low Clinical Pretest Probability and a d-dimer <1000(or equivalent), or with Moderate Clinical Pretest Probability and a D-dimer <500 (or equivalent) (e.g. suspected bleeding).
6. Ongoing need for anticoagulant therapy.
7. Suspected Pulmonary Embolism.
8. Superficial venous thrombosis that requires, or may require, anticoagulant therapy.
9. Life expectancy less than 3 months.
10. Previously confirmed episode of Deep Vein Thrombosis.
11. Geographic inaccessibility which precludes follow-up.
12. Known pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and females outpatients with a suspected Deep Vein Thrombosis
Sampling Method: Probability Sample
Enrollment: 1513 (Actual)
Dates: Start 2014-02; Primary Completion 2020-06-17 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Confirmed symptomatic proximal Deep Vein Thrombosis | within 90 days
  The primary outcome is confirmed symptomatic proximal Deep Vein Thrombosis (including involvement of the calf vein trifurcation but not isolated more distal Deep Vein Thrombosis; or pulmonary embolism (not including isolated sub-segmental abnormalities on Computed Tomography Pulmonary Angiogram; within 90 days (± 7 days for follow-up assessment) that is not diagnosed by scheduled diagnostic testing (includes events that occur between initial and scheduled follow-up proximal ultrasound examinations).

SECONDARY OUTCOMES:
Clinical Pretest Probability/ D-dimer/ Compression Ultrasound subgroups | within 90 days
  The primary outcome in the following subgroups:
  * Low Clinical Pretest Probability and D-dimer <1000 ug/L
  * Moderate Clinical Pretest Probability and D-dimer <500 ug/L
  * Moderate Clinical Pretest Probability and D-dimer 500 -999 ug/L
  * High Clinical Pretest Probability and D-dimer <500 ug/L
  * Low Clinical Pretest Probability and D-dimer 1000-2999 ug/L and negative initial ultrasound
  * Moderate Clinical Pretest Probability and D-dimer 1000-2999 ug/L and negative initial ultrasound
  * High Clinical Pretest Probability and D-dimer 500-1499 ug/L and negative initial ultrasound
Death | within 90 days
  Death within 90 days (± 7 days for follow-up assessment).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Levine, MD, Study Director — ocog
Locations (10):
- Canada (10):
  - University of Alberta Hospital, Edmonton, Alberta
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences - Hamilton General, Hamilton, Ontario
  - Hamilton Health Sciences - McMaster, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Juravinski Cancer Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital Regional Centre, Ottawa, Ontario
  - The Jewish General Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

REFERENCES:
- See also: Related Info — http://www.ocog.ca